CLINICAL TRIAL: NCT03968679
Title: Mapping of Sentinel Lymph Node Drainage Using SPECT/CT to Tailor Highly Selective Elective Nodal Irradiation in Node-negative Neck of Patients With Head and Neck Cancer
Brief Title: Lymph Drainage Mapping for Tailoring Elective Nodal Irradiation in Head and Neck Cancer
Acronym: SUSPECT-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M19SUS
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; lymph drainage mapping; sentinel node procedure; radiotherapy; unilateral elective neck irradiation
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unilateral elective nodal irradiation (Experimental): Exclusion of contralateral neck from elective nodal irradiation, based on results of SPECT/CT and (in case of contralateral drainage) contralateral sentinel node procedure.
  Interventions: Radiation: Unilateral elective nodal irradiation

INTERVENTIONS:
Radiation: Unilateral elective nodal irradiation — After injection of nanocolloid tracer submucosally around the tumor, patients undergo lymph drainage mapping (LDM) using SPECT/CT. If no contralateral drainage is visualized, the patient receives unilateral elective nodal irradiation (ENI). In case of contralateral lymph drainage, a contralateral sentinel node procedure is performed. If pathologic evaluation finds no metastasis, the patient receives unilateral ENI. If (micro/macro) metastasis are found, the patient will receive bilateral ENI.

SUMMARY:
This study aims to explore the safety and outcome of lymph drainage mapping(LDM) to individually tailor the elective nodal irradiation (ENI) to the ipsilateral neck only. The goal is to exclude the contralateral negative neck from the irradiation fields when there is no contralateral draining sentinel node. In case contralateral lymph drainage is found on SPECT/CT, a contralateral sentinel node procedure (SNP) is performed to remove the draining node. The patient will only receive contralateral ENI if (micro/macro)metastasis are found in this contralateral sentinel node.

DETAILED DESCRIPTION:
The SUSPECT2 study is a modified concept from the first SUSPECT study (N14SUS). The first study investigated whether lymph drainage mapping (LDM) using SPECT/CT was a safe and feasible method to exclude the contralateral neck from irradiation, or, in case of contralateral lymph drainage, to tailor the contralateral ENI field to the level containing the tracer accumulation. In this study, large dose reductions to most organs at risk were realized, as well as significant reductions of both short term (mucositis, dysphagia) and long term (xerostomia, dysphagia) toxicities.

Firstly, the SUSPECT2 study aims to expand the inclusion criteria of the original SUSPECT study. Secondly, it aims to further reduce the proportion of patients that undergoes bilateral ENI, by performing a contralateral sentinel node procedure (SNP) in case of contralateral lymph drainage. The patient will only receive contralateral ENI if (micro/macro)metastasis are found in this contralateral sentinel node.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and histopathologically proven primary HNSCC
* T1-4N0-2b
* Tumor does not cross midline
* WHO performance status 0 or 1
* Signed written informed consent

Exclusion Criteria:

* Distant metastatic spread at the time of inclusion
* Chemotherapy or surgery (for the present tumor), prior to inclusion
* Previous radiation treatment in the head and neck region, for any reason
* Previous neck dissection
* Recurrent or second primary tumor in the head and neck region
* Head and neck malignancies arising from skin, lip, nose, sinuses, nasopharynx, salivary glands, thyroid gland or esophagus
* Pregnancy or no active contraception for pre-menopausal women
* Known hypersensitivity to iodine or nanocolloid injection
* Having any condition (physical, mental, sociological) that interferes with the informed consent procedure and follow-up schedules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Contralateral regional failure | 1 year
  Cumulative incidence of contralateral regional metastasis.

SECONDARY OUTCOMES:
Treatment toxicity | Until 2 years after end of radiotherapy
  Physician-rated early and late treatment toxicity (CTCAE v5.0)
Health-related quality of life | Until 18 months after end of radiotherapy
  Health-related quality of life after treatment (EORTC QLQ-C30/HN35)

CONTACTS AND LOCATIONS:
Overall Officials: Abrahim Al-Mamgani, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Veij Mestdagh PD, Schreuder WH, Vogel WV, Donswijk ML, van Werkhoven E, van der Wal JE, Dirven R, Karakullukcu B, Sonke JJ, van den Brekel MWM, Marijnen CAM, Al-Mamgani A. Mapping of sentinel lymph node drainage using SPECT/CT to tailor elective nodal irradiation in head and neck cancer patients (SUSPECT-2): a single-center prospective trial. BMC Cancer. 2019 Nov 14;19(1):1110. doi: 10.1186/s12885-019-6331-8. PMID 31727019